CLINICAL TRIAL: NCT07084857
Title: "Association Between Isokinetic Lower Extremity Muscle Strength and Bone Mineral Density in Elderly Women With and Without Osteoporosis: A Case-Control Study"
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azza Mohammed, Prof. Dr, Cairo University
Other Study IDs: Faculty of Physical Therapy CU; faculty of physical therapy (Registry Identifier: faculty of physical therapy)
Record Dates: First submitted 2025-05-20; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bone Mineral Density; Isokinetic Strength; Hip Muscles; Knee Muscles; Elderly Women
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: correlational analysis between BMD and isokinetic lower extremity strength — correlational analysis between BMD and isokinetic lower extremity strength

SUMMARY:
bone density and muscle strength appear to be more related to each other. Examining the association between muscle strength and bone health is very important in recognizing risk factors for lower extremity muscle weakness.

DETAILED DESCRIPTION:
Dual Energy X-ray Absorptiometry (DEXA) scan will be used to assess hip bone mineral density (BMD) at femoral head region. Isokinetic PT of hip flexors, extensors, abductors and adductors and knee flexors and extensors will be measured using Biodex System 3 Isokinetic Dynamometer. The measured outcomes will be evaluated at an angular velocity of 60°/sec in a concentric mode of muscle contraction for five successive repetitions. Isokinetic testing will be done at the Isokinetic Laboratory, Faculty of Physical therapy, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

1. The group of OP (n=33) has femoral BMD T-scores below -2.5 diagnosed by DEXA scan according to the WHO [8] classification of BMD in 2003,
2. The control group has normal BMD T-scores more than -1.

Exclusion Criteria:

1. There was any neurological, musculoskeletal, rheumatologic, respiratory or cardiovascular problem.
2. They were receiving medications that result in bone loss such as corticosteroids,
3. They had vertigo, dizziness, or any vestibular problem,
4. They had hyperthyroidism or hyperparathyroidism. 6- They actively participate in sports activities,
5. They underwent previous surgery (e.g; joint replacement) or history of fractures of the lower extremity.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on a sample size calculation via G Power software, a total of 70 participants will be required to participate in the study taking in consideration 20% drop out. A total 66 elderly women with ages range from 50 to 70 years will be involved in the study
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
isokinetic strength of hip muscles | one month
  isokinetic hip muscle stregth will be measured using Biodex system 3 Isokinetic Dynamometer
Bone mineral density | one month
  bone mineral density measured by dual energy x ray absorptiometry scan

SECONDARY OUTCOMES:
isokinetic strength of knee muscles | one month
  isokinetic hip muscle stregth will be measured using Biodex system 3 Isokinetic Dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Azza Mohammed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided